CLINICAL TRIAL: NCT01411111
Title: An Open Label, Sequential, Single Cohort, Repeat Dose Study to Investigate the Potential Interaction of GSK2190915 on the Pharmacokinetics of Rosuvastatin in Healthy Adult Subjects.
Brief Title: A Repeat Dose Study to Investigate the Interaction of GSK2190915 on the Pharmacokinetics of Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112362
Record Dates: First submitted 2011-04-14; First posted 2011-08-08 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: Drug-drug interaction; rosuvastatin; asthma; FLAP inhibitor
MeSH Terms: conditions — Asthma | interventions — Rosuvastatin Calcium; 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin foll by GSK2190915 30mg + rosuvastatin (Active Comparator): Subjects will be orally administered rosuvastatin 10 mg/day for 7 days in treatment period 1. The subjects will then receive rosuvastatin 10 mg/day in combination with GSK2190915 30 mg/day for 7 days in treatment period 2A.
  Interventions: Drug: Rosuvastatin 10 mg; Drug: GSK2190915 30mg
- Rosuvastatin foll by GSK2190915 100mg + rosuvastatin (Active Comparator): Subjects will be orally administered rosuvastatin 10 mg/day for 7 days in treatment period 1. The subjects will then receive rosuvastatin 10 mg/day in combination with GSK2190915 100 mg/day for 7 days in treatment period 2B.
  Interventions: Drug: Rosuvastatin 10 mg; Drug: GSK2190915 100mg

INTERVENTIONS:
Drug: Rosuvastatin 10 mg — days 1-14
Drug: GSK2190915 30mg — 1x30mg tablet, days 8-14
  Arms: Rosuvastatin foll by GSK2190915 30mg + rosuvastatin
Drug: GSK2190915 100mg — 1x100mg tablet, days 8-14
  Arms: Rosuvastatin foll by GSK2190915 100mg + rosuvastatin

SUMMARY:
Leukotrienes are potent inflammatory molecules produced mainly by mast cells, eosinophils, monocytes/macrophage and neutrophils in response to allergic or inflammatory stimuli. GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor that attenuates the production of leukotrienes, through the blockage of the first committed step in the leukotriene pathway, 5 lipoxygenase (5-LO) activation.

GSK2190915 has been shown to be an in vitro inhibitor of human organic anion transporting polypeptides 1B1 and 1B3 (OATP1B1 and OATP1B3), hence there is a potential for a pharmacokinetic drug-drug interaction with OATP1/ B1 substrates such as the anti-lipidemic rosuvastatin.

This study will evaluate the effect of repeat oral dosing of GSK2190915 (30milligram (mg) and 100mg) on the steady-state pharmacokinetics (PK) of rosuvastatin (10 mg). In addition, the study will evaluate the safety and tolerability of this combination when co-administered to healthy, adult volunteers in two cohorts.

DETAILED DESCRIPTION:
GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor that attenuates the production of leukotrienes, through the blockage of the first committed step in the leukotriene pathway, 5 lipoxygenase (5-LO) activation. Leukotrienes are potent inflammatory molecules produced mainly by mast cells, eosinophils, monocytes/macrophage and neutrophils in response to allergic or inflammatory stimuli. As GSK2190915 inhibits the production of leukotriene B4 and cysteinyl leukotrienes it has strong potential utility in the treatment of asthma and Chronic Obstructive Pulmonary Disease (COPD) The organic anion transporting polypeptides (OATP's) form a superfamily of sodium-independent transport systems that mediate the transmembrane transport of a wide range of amphipathic organic compounds. Of the 11 human OATP transporters, OATP1B1, and OATP1B3 are specifically expressed on the sinusoidal membrane of hepatocytes and are considered to be of particular importance for hepatic drug elimination and drug pharmacokinetics.

GSK2190915 has been shown to be an inhibitor of OATP1B1 and OATP1B3. Several clinically utilised drugs have been identified as substrates of OATP transporters, including rosuvastatin - a member of the statin group of anti-lipidemics.

As the target patient population for GSK2190915 may overlap with that for statins such as rosuvastatin, it is important to evaluate any potential effects of GSK2190915 on the pharmacokinetics of a statin known to undergo hepatic elimination via OATP1B1/1B3 This study will evaluate the effect of repeat oral dosing of GSK2190915 on the steady-state pharmacokinetics of rosuvastatin. In addition, the study will evaluate the safety and tolerability of this combination when co-administered to healthy, adult volunteers.

Two dose levels of GSK2190915 will be investigated; 30mg and 100mg once daily for 7 days. The rosuvastatin dose selected for this study is 10mg which allows for up to a 4 times increase in systemic exposure if there is a pharmacokinetic interaction.

The study will be an open label, single-sequence study in two cohorts with 2 treatment periods. 28 subjects will receive rosuvastatin 10mg/day for 7 days during the first treatment period, following on from which 14 subjects each will receive either GSK2190915 30 mg/day or GSK2190915 100mg/day in combination with rosuvastatin 10mg/day for the next 7 days. Subjects will be followed up 7-14 days after their last dose. PK samples will be obtained for both rosuvastatin and GSK2190915 during the study. Safety will be evaluated via physical examinations, ElectroCardioGrams (ECG) and vital signs.

Approximately 28 healthy subjects will be enrolled such that approximately 24 subjects (12 in each of the two treatment arms) complete dosing and critical assessments.

ELIGIBILITY:
Inclusion Criteria:

* The subject is of non-Asian origin.
* Aspartate aminotransferase (AST), Alanine aminotransferase (AMT), alkaline phosphatase and bilirubin <1.5xULN (upper limit of normal) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination and laboratory tests. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included if the Investigator believes that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. The GSK medical monitor will be consulted where necessary.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.

  • A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 Milli lnternational Units/millilitre ( MIU/ml) and estradiol < 40 picogram/ml (pg/ml) (<147 picomoles/Litre (pmol/L)) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 or the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment. For most forms of HRT, at least 2- 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Body weight ≥ 50 kilograms (kg) (110 lbs) for men and ≥ 45 kg (99lbs) for women and BMI (body mass index) within the range 18-30 kg/m2 inclusive.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* 12 lead ECG (electrocardiogram) without any clinically significant abnormality as judged by the Investigator, and average QTc (corrected QT duration), QTcB or QTcF < 450 msec

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Current, or history of, muscle complaints (e.g. unexplained weakness, tenderness, pain), myopathy or rhabdomyolysis.
* Current, or history of, renal impairment or insufficiency.
* Current, or history of, hypothyroidism.
* Lactose intolerant, including galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* A positive pre-study drug/alcohol screen.
* A positive test for HIV (Human Immunodeficiency Virus) antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Pregnant females as determined by positive serum hCG (Human chorionic gonadotrophin) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels or breath CO levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01-06 (Actual); Primary Completion 2011-02-23 (Actual); Study Completion 2011-02-23 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) of rosuvastatin | On 7 and 14 days post- first dose
Area Under the Curve(0-τ) of rosuvastatin | On 7 and 14 days post first dose

SECONDARY OUTCOMES:
Safety and tolerability as assessed by clinical monitoring of blood pressure, pulse rate, ECG monitoring and laboratory safety data, as well as reporting of Adverse Events in healthy adult subjects from dosing to one week post-dose. | From screening to follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112362 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112362?search=study&search_terms=112362#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register